CLINICAL TRIAL: NCT01893437
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Single Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO6799477 Following Oral Administration of Single Ascending Doses in Healthy Volunteers.
Brief Title: A Study of RO6799477 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP28751; 2013-000402-28 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Single oral dose group (Experimental)
  Interventions: Drug: RO6799477

INTERVENTIONS:
Drug: RO6799477 — Single doses of RO6799477

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled, single dose study will investigate the safety, pharmacokinetics, pharmacodynamics of RO6799477 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers, aged 18-45 years, inclusive
* Male volunteers with female partner of childbearing potential must agree to use an effective form of birth control during the study and for 3 months after discontinuation of treatment.
* Body Mass index (BMI) of 18-30 kg/m2, inclusive

Exclusion Criteria:

* Infection with human immunodeficiency virus antibody (HIV 1 and 2), Hepatitis B, hepatitis C
* Positive testing for drugs of abuse
* Any history of alcohol and/or drug of abuse addiction

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety: Incidence of adverse events | 18 weeks

SECONDARY OUTCOMES:
Part 1 and 2: Pharmacokinetics: plasma concentration of RO6799477 | Pre-dose, Day 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leiden, Netherlands